CLINICAL TRIAL: NCT03903042
Title: Comparison of Aurora Fundus Camera With Traditional Fundus Camera in Diabetic Retinopathy With Phoebus Visual Artificial Intelligence
Brief Title: Comparison of Aurora Fundus Camera With Traditional Camera in Diabetic Retinopathy With Visual Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Fenghua Wang, Doctoral Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Shanghai1stAI
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Retinopathy
Keywords: Aurora fundus camera; Artificial intelligence; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Center 1: Traditional camera(Canon) vs Aurora camera
- Group 2: Center 2: Traditional camera(Zeiss) vs Aurora camera
- Group 3: Center 3: Traditional camera(Topcon) vs Aurora camera

SUMMARY:
This study aims to compare the effect of Aurora handheld fundus camera with traditional desktop fundus camera in the fundus photography screening of diabetic patients, and to evaluate the effect of artificial intelligence algorithm in the diagnosis of diabetic retinopathy.

DETAILED DESCRIPTION:
Aurora handheld fundus cameras are used to take fundus photography on diabetic patients in 3 ophthalmic diabetic retinopathy screening centers in China to compare its effect with the hospital's traditional desktop fundus camera, and evaluate the auxiliary diagnostic effect of Phoebus artificial intelligence algorithm in diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are more than 18 years of age, male or female Chinese patients;
2. Diagnosed with diabetes;
3. Prior written informed consent should be obtained

Exclusion Criteria:

1. Patients with invisible fundus caused by any cause;
2. Patients or his/her licensor unwill to sign an informed consent or follow this protocol;
3. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with diabetes, more than 18 years of age, male or female Chinese patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Image Quality of Aurora camera | within 3 months
  Score of Image Quality

SECONDARY OUTCOMES:
Outcome of gold standard | within 3 months
  Gold standard: 8 photographs of one patient(4 by Aurora camera, 4 by traditional camera) by ophthalmologist（double blinded）
Image of Aurora camera | 1 month
  Images taken by Aurora camera
Image of traditional camera (Center 1: Canon) | 1 month
  Image taken by traditional camera（Center 1: Canon, pupil not dilated）
Image of traditional camera (Center 2: Zeiss) | 1 month
  Image taken by traditional camera（Center 2: Zeiss, pupil dilated）
Image of traditional camera (Center 3: Topcon) | 1 month
  Image taken by traditional camera（Center 3: Topcon, pupil dilated）
Outcome of artificial intelligence algorithm | 3 months
  Outcome of artificial intelligence algorithm(Normal or Referral Required)

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Wang, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report will be published
Supporting Information: CSR
Time Frame: starting 6 months after publication
Access Criteria: Dr Fenghua Wang will review requests and criteria.

REFERENCES:
- [Background] Jin G, Xiao W, Ding X, Xu X, An L, Congdon N, Zhao J, He M. Prevalence of and Risk Factors for Diabetic Retinopathy in a Rural Chinese Population: The Yangxi Eye Study. Invest Ophthalmol Vis Sci. 2018 Oct 1;59(12):5067-5073. doi: 10.1167/iovs.18-24280. PMID 30357401
- [Background] Zheng X, Zhang L. A study of retinopathy analysis in type 2 diabetes patients in Chinese population. Pak J Pharm Sci. 2018 Sep;31(5(Supplementary)):2041-2046. PMID 30393210
- [Background] Hendrick AM, Gibson MV, Kulshreshtha A. Diabetic Retinopathy. Prim Care. 2015 Sep;42(3):451-64. doi: 10.1016/j.pop.2015.05.005. PMID 26319349
- [Background] Wong TY, Bressler NM. Artificial Intelligence With Deep Learning Technology Looks Into Diabetic Retinopathy Screening. JAMA. 2016 Dec 13;316(22):2366-2367. doi: 10.1001/jama.2016.17563. No abstract available. PMID 27898977
- [Background] Abramoff MD, Niemeijer M, Russell SR. Automated detection of diabetic retinopathy: barriers to translation into clinical practice. Expert Rev Med Devices. 2010 Mar;7(2):287-96. doi: 10.1586/erd.09.76. PMID 20214432
- [Background] Li Z, Keel S, Liu C, He Y, Meng W, Scheetz J, Lee PY, Shaw J, Ting D, Wong TY, Taylor H, Chang R, He M. An Automated Grading System for Detection of Vision-Threatening Referable Diabetic Retinopathy on the Basis of Color Fundus Photographs. Diabetes Care. 2018 Dec;41(12):2509-2516. doi: 10.2337/dc18-0147. Epub 2018 Oct 1. PMID 30275284